CLINICAL TRIAL: NCT02626676
Title: Nutrition Educational Programme Impact on Serum Phosphate Control
Brief Title: Educational Programme Impact on Serum Phosphate Control
Acronym: EPIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcus Vinicius de Souza Joao Luiz, MSC., Pharm.D., University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USAoPaulo EPIC
Record Dates: First submitted 2015-12-06; First posted 2015-12-10 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Renal Insufficiency, Chronic
Keywords: renal dialysis, hyperphosphatemia, educational programme
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Educational Programme Group (Experimental): Stage 5D Chronic Kidney Disease Patients on high-efficiency hemodialysis programme - 4-hour sessions, 3 times a week will be followed up
  Interventions: Other: Educational Programme

INTERVENTIONS:
Other: Educational Programme — Educational Programme consists of lectures and group dynamics about nutrition during hemodialysis sessions.

SUMMARY:
Background: In Chronic Kidney Disease patients, it is crucial to begin treatment as soon as possible in order to minimize the complication-related risks. Encouraging patients to adhere to their treatment plans is a great challenge for health care professionals. Objectives: The aim of this study is to evaluate the impact of a nutrition educational programme on the hyperphosphatemia using the transtheoretical model of eating behavior. Subjects and Methods: A prospective Interventional study is being conducted in a dialysis centre with 180 stage 5D Chronic Kidney Disease patients who exhibit phosphate serum levels > 5.5 mg/dL. The educational intervention consists of lectures and group dynamics sessions performed during dialysis sessions. Anthropometric, clinical, demographic and laboratory parameters (serum phosphorus concentration will be evaluated and the transtheoretical model of eating behavior (TMFB) will be applied pre- and post-intervention.

DETAILED DESCRIPTION:
Background: In Chronic Kidney Disease patients, it is crucial to begin treatment as soon as possible in order to minimize the complication-related risks. Encouraging patients to adhere to their treatment plans is a great challenge for health care professionals. Objectives: The aim of this study is to evaluate the impact of a nutrition educational programme on the hyperphosphatemia using the transtheoretical model of eating behavior. Subjects and Methods: A prospective Interventional study is being conducted in a dialysis centre with 180 stage 5D Chronic Kidney Disease patients who exhibit phosphate serum levels > 5.5 mg/dL. The educational intervention consists of lectures and group dynamics sessions performed during dialysis sessions. Anthropometric (weight, height, body mass index), clinical, demographic (sex, age, time on dialysis programme, literacy/schooling) and laboratory parameters (phosphate serum levels) will be evaluated and the transtheoretical model of eating behavior (TMFB) will be applied pre- and post-intervention. Reduction of phosphate serum levels and positive/negative behavioral changes will be the evaluated outcomes. Statistical Analyses will be carried out in order to compare the effect of educational programme on phosphate serum levels and on the behaviour changes.

ELIGIBILITY:
Inclusion Criteria:

* patients who freely consent to participate in this study
* aged from 18 years or older
* both genders
* phosphate serum levels higher than 5.5 mg/dl (last 3 consecutive monthly measures)

Exclusion Criteria:

* patients who do not consent to participate in this study
* pregnant
* cognitive deficit
* mental diseases
* patients whose phosphate serum levels lower than 5.5 mg/dl or equal to 5.5 mg/dl

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Reduction of PhosphateSerum Level | 3 months
  Phosphate Serum Levels above or equal 5.5 mg/dl will be monitored in order to identify reduction

SECONDARY OUTCOMES:
Positive or Negative Behavioral Change According to the Transtheoretical Model of Eating Behavior | 3 months
  After intervention (3 months), it will be identified whether patients show Positive or Negative Behavioral change (according to the transtheoretical model of eating behavior) will be identified

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Vinicius SJ LUIZ, MSc, PharmD, Principal Investigator — University of Sao Paulo
Locations (1):
- RenalClass, Dialysis Centre, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No